CLINICAL TRIAL: NCT03866317
Title: A Pilot Study to Assess the Safety and Efficacy of Secukinumab in Alleviating Symptoms of Discoid Lupus Erythematosus
Brief Title: A Study to Assess the Safety and Efficacy of Secukinumab in Alleviating Symptoms of Discoid Lupus Erythematosus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting participants
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Gideon Piers Smith, Vice Chair, Department of Dermatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000403
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Discoid Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — secukinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Secukinumab (Experimental): Secukinumab 300 mg injection at week 0, 1, 2, 3, 4, then every 4 weeks until week 12
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — All subjects will receive secukinumab 300 mg injections subcutaneously at week 0, 1, 2, 3, 4, then every 4 weeks until week 12.
  Other Names: Cosentyx

SUMMARY:
Discoid lupus erythematosus is a chronic inflammatory skin condition and may lead to itch, skin pain, open sores, scarring, disfigurement and hair loss. Studies have shown that IL-17A may play a major role in inflammation and in the pathogenesis of discoid lupus. Treatment of discoid lupus sometimes is a challenge and unresponsive to current therapies. Secukinumab, an anti-IL-17A monoclonal antibody has been safe and effective in the treatment of psoriasis. The investigators propose to study the efficacy and safety of secukinumab in discoid lupus.

DETAILED DESCRIPTION:
Discoid lupus erythematosus (DLE) is a cutaneous manifestation of lupus that can exist either as part of systemic lupus erythematosus (SLE), or as a chronic cutaneous condition with no systemic involvement. While the skin-limited, chronic form, has no impact on mortality, it can have significant morbidity, as lesions are painful and scarring. While some patients respond well to use of steroids, whether topical or intralesional, antimalarials such as hydroxychloroquine, or traditional immuno-suppressants there is a significant proportion of patients who remain non-responsive to these treatments, or require high dosages of these, oral steroids, or experimental therapies to suppress the condition. For this group of patients there is a high clinical need to find alternate therapies.

Although the pathways of inflammation are poorly understood, one cytokine of potential interest is IL-17A. Immunohistochemical analysis of skin samples from 89 subjects showed that expression of IL-17A was higher in DLE, SCLE and SLE patients than in negative control subjects (all p<0.05). Serum IL-17A concentrations were higher in DLE and SLE patients than in negative controls (p<0.05), a finding confirmed in studies of DLE in different populations.

Recently secukinumab (Cosentyx), an anti-IL-17A monoclonal antibody, has been approved for use in psoriasis after rapid and sustained results in clinical trials. It has also found promise in other inflammatory conditions where IL-17A signaling is believed to be important, such as uveitis.

Given its good safety profile, its impressive response in psoriasis and steroid-unresponsive inflammatory conditions, and the immunohistochemical evidence that IL-17A may be important in the inflammatory path of DLE, the investigators propose a pilot study of secukinumab in discoid lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18 years of age or older
2. Subjects with moderate to severe DLE with at least one active discoid target lesion (0.5-1.0 cm2), with CLASI ≥ 5.
3. Willingness of subject to follow all study procedures
4. Willingness to avoid excessive exposure of diseased areas to natural or artificial sunlight

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Any condition or therapy that in the investigator's opinion may pose a risk to the subject or that could interfere with any evaluation in the study
3. Systemic Lupus Erythematosus (SLE) as defined by ACR criteria
4. Known hypersensitivity to any of the constituents or excipients of the investigational product
5. Use of any prescription or non-prescription medication that could interfere with efficacy evaluations in the study
6. Change in use of systemic DLE therapy, e.g. systemic corticosteroids, cyclosporine A, azathioprine, mycophenolate mofetil, in the past 1 month.
7. Use of systemic pain medications, e.g. oxycodone in the past 2 weeks
8. Participation in another clinical research study with an investigational drug within 4 weeks before this study
9. Use of immune-suppressant or other biological treatment
10. Starting antimalarial medicine after enrolling in the study. Subjects who are already on a stable dose of antimalarial before enrollment, may continue the same dose.
11. An ongoing infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of Secukinumab in Discoid Lupus Erythematosus by clinical responder rate at week 16. | 16 week
  By using the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Smith, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- CURTIS (Massachusetts General Hospital), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided